CLINICAL TRIAL: NCT01565161
Title: Healthy Habits, Happy Homes: An Intervention to Improve Household Routines for Obesity Prevention
Acronym: HH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Elsie Taveras, Associate Professor, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: U48 DP001946-5033375; U48DP001946 (NIH)
Record Dates: First submitted 2012-03-26; First posted 2012-03-28 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Obesity
Keywords: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Home-Based Health Coaching (Experimental): Intervention delivered in the home.
  Interventions: Behavioral: Home-Based Health Coaching
- Control Arm (Active Comparator): Mailed educational materials
  Interventions: Behavioral: Mailed materials

INTERVENTIONS:
Behavioral: Home-Based Health Coaching — The 6-month intervention arm consists of 3 components:
  1. In-home coaching visits with a health educator trained in motivational interviewing to encourage behavior change. In addition to 4 monthly in-home coaching visits, participants receive 4 monthly coaching phone calls to supplement the in-person visits.
  2. Use of mobile technology to deliver health information by text message - participants receive messages twice weekly for 16 weeks and then weekly for 8 weeks of the program. Those without a phone capable of receiving text messages receive postcards by mail.
  3. Printed materials, including educational handouts, newsletters, and activities highlighting target behaviors, sent monthly for 4 months.
  Other Names: Healthy Habits, Happy Homes Health Coaching
  Arms: Home-Based Health Coaching
Behavioral: Mailed materials — We designed materials for our control group focusing on Developmental milestones during early childhood to provide information that participants would find relevant and helpful for parenting, but that would also not influence intervention behaviors, such as TV viewing or household routines related to sleeping, eating, or television viewing.
  Participants received 4 monthly mailing packages, each focusing thematically on one of four milestone domains: motor, language, cognitive and social/emotional. Educational materials were adapted from the Center for Disease Control's "Positive Parenting Tips for Healthy Child Development", and the mailing included child-appropriate incentives to reinforce the concepts presented in the educational materials.
  Other Names: Healthy Habits, Happy Homes mailed materials
  Arms: Control Arm

SUMMARY:
While childhood obesity rates may have plateaued in some US population subgroups, such as whites and those of higher socioeconomic status, overall rates of obesity remain high and racial/ethnic and socioeconomic disparities appear to be widening. Among the most promising approaches for childhood obesity prevention and management are interventions that begin early in life and that support change at the individual and community levels.

The goal of this project is to develop and test an intervention delivered to racial/ethnic minority and low income parents of 2-5 year old children in their homes, designed to promote adoption of household routines and parenting strategies that are preventive of obesity. To achieve this goal, the investigators will work with community health centers in Boston, Cambridge, and Somerville to recruit families to participate in an individual-level randomized controlled trial. The investigators partner community health centers include the Roxbury Comprehensive Community Health Center, Dimock Community Health Centers, and the Cambridge Health Alliance (CHA).

Participants will be randomized to receive either 1) mailed educational materials for the duration of the 6-month program (control), or 2) home-based health coaching visits and phone calls with a health educator, text messages, and educational materials promoting the adoption of household routines and target behaviors (intervention).

The investigators goal is to evaluate the feasibility and effectiveness of the investigators designed intervention (as compared to the control condition) using baseline and post-intervention data. In order to do so, the investigators will assess change from baseline to post-intervention in the investigators key behavioral outcomes of interest, including adoption of three household routines:

1. Regularly eating meals together as a family
2. Obtaining adequate sleep
3. Limiting screen-viewing time

ELIGIBILITY:
Inclusion Criteria:

* Parent with child between 2-5 years old
* Child has a TV in the room where s/he sleeps
* Parent is comfortable reading, writing and having conversations in English or Spanish
* Child was seen for a well-child care visit at one of collaborating community health centers in the last 90 days

Exclusion Criteria:

* Parent is not 18 years or older
* Family is planning to move from the Boston area in the net 6 months
* Child has a physical/mental health condition which requires chronic care

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 117 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Parent and child health behaviors | Baseline, 6 months
  Using parent self-report surveys, we will assess change from baseline to post-intervention in parent and child behaviors related to the following health outcomes:
  * TV viewing, including TV in the room where the child sleeps, time spent watching TV, total screen time
  * Sleep, including parent and child sleep duration and presence of a calming nighttime routine
  * Diet, including eating meals together as a family, lowering intake of fast food, and lowering intake of sugar-sweetened beverages
TV Viewing Time | Baseline, 6 months
  Using two separate measures of Child TV viewing time (parent-report and measured TV time using the TV Allowance device, we will assess change from baseline to post-intervention in the amount of TV the child watches.
  Additionally, using parent-report surveys we will assess change from baseline to post-intervention in total screen time as well as observed presence of TV in the room where the child sleeps.

SECONDARY OUTCOMES:
Child height and weight measurements | Baseline, 6 months
  We will assess change in child BMI and BMI z-score from baseline to post-intervention using in-person child height and weight measurements, taken by trained research staff using a standing Schorr board to measure height and an electronic scale to measure weight.
Cognitive stimulation in the home | Baseline, 6 months
  We will assess change from baseline to post-intervention in total score on the STIMQ, a validated instrument that captures the presence of cognitive stimulation in the home. This instrument is administered as an in-person interview with the primary caregiver.
Presence of media devices in the home | Baseline, 6 months
  We will assess the home environment at baseline and post-intervention, using a developed instrument called the Home Environment Media Inventory (HEMI). From this, we will be able to observe change from baseline to follow up in the presence of media devices in the home, as well as basic neighborhood and household characteristics. Media devices measured include: TV, DVD, DVR/Tivo, Cable, and Computer.
Use of mobile technology | Baseline
  We will assess the participant's use of mobile technology at baseline, such as text messaging and downloaded applications, as well as whether participants have had their cell service cut off for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care; Julia McDonald, MS, MPH, Study Director — Harvard Pilgrim Health Care
Locations (2):
- Harvard Pilgrim Health Care, Boston, Massachusetts, United States
- University of Guelph, Guelph, Ontario, Canada

REFERENCES:
- [Derived] Sharifi M, Dryden EM, Horan CM, Price S, Marshall R, Hacker K, Finkelstein JA, Taveras EM. Leveraging text messaging and mobile technology to support pediatric obesity-related behavior change: a qualitative study using parent focus groups and interviews. J Med Internet Res. 2013 Dec 6;15(12):e272. doi: 10.2196/jmir.2780. PMID 24317406
- [Derived] Haines J, McDonald J, O'Brien A, Sherry B, Bottino CJ, Schmidt ME, Taveras EM. Healthy Habits, Happy Homes: randomized trial to improve household routines for obesity prevention among preschool-aged children. JAMA Pediatr. 2013 Nov;167(11):1072-9. doi: 10.1001/jamapediatrics.2013.2356. PMID 24019074
- [Derived] Taveras EM, McDonald J, O'Brien A, Haines J, Sherry B, Bottino CJ, Troncoso K, Schmidt ME, Koziol R. Healthy Habits, Happy Homes: methods and baseline data of a randomized controlled trial to improve household routines for obesity prevention. Prev Med. 2012 Nov;55(5):418-26. doi: 10.1016/j.ypmed.2012.08.016. Epub 2012 Aug 30. PMID 22960162